CLINICAL TRIAL: NCT05914610
Title: Envollizumab Combined With Fruquintinib and SOX Versus SOX for Conversion Therapy in Her-2 Negative Unresectable Locally Advanced Gastric Cancer: a National Multicenter Randomized Controlled Study
Brief Title: Envollizumab Combined With Fruquintinib and SOX Versus SOX for Conversion Therapy in Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Clinical Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-028
Record Dates: First submitted 2023-05-27; First posted 2023-06-22 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — HMPL-013; Oxaliplatin; Tegafur

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Envolimab + fruquinitinib +SOX regimen (Experimental)
  Interventions: Drug: Envolimab; Drug: Fruquintinib; Drug: Oxaliplatin; Drug: Tegafur
- SOX regimen (Active Comparator)
  Interventions: Drug: Oxaliplatin; Drug: Tegafur

INTERVENTIONS:
Drug: Envolimab — Envolizumab 300mg, D1, ih, Q3W 4-6cycles
  Arms: Envolimab + fruquinitinib +SOX regimen
Drug: Fruquintinib — Fruquinitinib 3mg/d, QD, PO, D1-D14, Q3W 4-6cycles
  Arms: Envolimab + fruquinitinib +SOX regimen
Drug: Oxaliplatin — Oxaliplatin 130 mg/m2, ivgtt 0-2h, D1, Q3W 4-6cycles
Drug: Tegafur — Tegafur was calculated according to body surface area , P.O., bid, d1-d14#And the dosage according body surface area:<1.25m2, 40mg every time;1.25-1.5m2,50mg every time; >1.5m2, 60mg every time Q3W 4-6cycles

SUMMARY:
To investigate the clinical efficacy and safety of envollizumab combined with fruquintinib and SOX versus SOX in conversion therapy for patients with Her-2 negative, unresectable locally advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years of age;
2. Pathological (including histological or cytological) confirmation of gastric adenocarcinoma;
3. Before surgery, CT/MRI, PET-CT, if necessary, laparoscopic exploration to determine the clinical stage of T4bN0M0 and TanyN2-3M0, and determined by researchers that the local advanced patients can not be resectable;
4. At least one measurable detected by CT examination in accordance with the RECIST1.1
5. ECOG#Eastern Cooperative Oncology Group#PS#Performance Status#:0-1 scores;
6. The expected survival time is more than 3 months
7. The main organ function is normal, which should meet the following criteria:

   #1#blood routine examination standards should be met#no blood transfusion within 14 days#

   a.HB≥ 100g/L b. WBC≥3×109/L c. ANC≥1.5×109/L d. PLT≥100×109/L #2#biochemical examination shall comply with the following criteria#
   1. BIL#1.5 normal upper limit ULN
   2. ALT and AST#2.5 ULN
   3. Cr≤1 ULN#CCR#creatinine clearance rate##60ml/min(Cockcroft Gault formula)
8. Women of childbearing age must have a pregnancy test in 7 days before entering the group (in serum), and the results were negative, and willing to use appropriate contraception during the study period and the last 8 weeks after giving drug test; men should have the surgical sterilization, or adopt the appropriate contraceptive methods during the test and the last 8 weeks after giving drug test#
9. No other clinical studies were conducted before and during the treatment
10. Participants is willing to participate in this study, sign the informed consent, have good compliance, cooperate with follow-up

Exclusion Criteria:

1. Imaging or intraoperative exploration found patients with peritoneum, liver, lung and other distant metastases
2. Patients with allergies or suspected allergies to study drugs or similar drugs
3. Confirmed HER-2 positive patients
4. Other malignancies in the past 5 years, except basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix
5. Live vaccine was administered within 4 weeks prior to enrolling or possibly during the study period
6. Had an active autoimmune disease or a history of autoimmune disease within 4 weeks prior to enrollment
7. Past recipients of allogeneic bone marrow transplants or organ transplants
8. Patient has any current disease or condition that affects drug absorption, or the patient is unable to take the drug orally
9. The blood pressure of patients with hypertension cannot be reduced to the normal range by the one antihypertensive drugs (systolic pressure ≥150 mmHg, diastolic pressure ≥100 mmHg) or hard to controled by two or more antihypertensive drugs
10. Patients are positive of urine protein (urine protein detection 2+ or above, or 24 hours urine protein quantitative >1.0g)
11. The patient currently has gastrointestinal diseases such as active gastric and duodenal ulcers, ulcerative colitis, or active bleeding from unresectosed tumors, or other conditions determined by researchers that may cause gastrointestinal bleeding or perforation
12. Patients with significant evidence or history of bleeding tendency within 3 months prior to enrollment (bleeding within 3 months >30 mL, hematemesis, black stool, blood in stool), hemoptysis (within 4 weeks >5 mL fresh blood) or a thromboembolic event (including stroke and/or transient ischemic attack) within 12 months
13. Cardiovascular disease of significant clinical significance, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within 6 months prior to enrollment; New York Heart Association (NYHA) Grades for Congestive Heart Failure more than class II ; Ventricular arrhythmias requiring medical treatment; An electrocardiogram (ECG) showed a QT c interval ≥480 milliseconds
14. Active or uncontrolled severe infection (≥CTCAE grade 2 infection)
15. A history of human immunodeficiency virus (HIV) infection or clinically significant liver disease, including viral hepatitis [active HBV infection must be ruled out as a known carrier of hepatitis B virus (HBV), i.e. positive HBV DNA (>1×104 copies /mL or >2000 IU/ml); known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL), or other hepatitis, cirrhosis]
16. The researchers consider those who were not suitable for inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Surgical conversion rate | 2-3 months
  Defined as the proportion of patients who have undergone surgical resection after multidisciplinary assessment after completing 4-6 cycles of conversion therapy

SECONDARY OUTCOMES:
Pathological complete response (pCR) | 4 months
  Measured as the proportion of participants with a pathological complete response at the time of definitive surgery.
Median disease free survival (DFS) time | 3 years
  The time from opreation to the time when only 50% of the individuals had no relapse or tumor progression
1-year DFS rate | 1 year
3-year DFS rate | 3 years
Objective response rate (ORR) | 4 months
  Defined as the percentage of the participants in the analysis population who had a confirmed patial response and complete reponse according to RECIST 1.1 based on investigator assessment
Major pathological response rate (MPR) | 4 months
  The proportion of participants with a major pathological response (mPR) at the time of definitive surgery.
R0 resection rate | 2-3 month
  Defined as no residue under the microscope after resection
Median survival time | 3 years
  The time from enrollment to the time when only 50% of the individuals alive
Adverse event (AEs) | 2 years
  Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. The number of Participants with adverse events will be recorded at each treatment visit.
Quality of life (QOL) | 2 years
  The quality of life of patients during treatment is eveluated by the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 (V3.0)